CLINICAL TRIAL: NCT07232108
Title: Effects of Intrathecal Morphine Compared With Trocar-Site Infiltration and Intraperitoneal Bupivacaine on Postoperative Quality of Recovery and Inflammatory Markers After Laparoscopic Hysterectomy: A Prospective, Randomized, Double-Blind Controlled Trial
Brief Title: Intrathecal Morphine Versus Trocar-Site and Intraperitoneal Bupivacaine for Quality of Recovery After Laparoscopic Hysterectomy
Acronym: ITM-LH-QoR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Principal Investigator Ayşenur Dostbil, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/697; 2025/1 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain Management; Laparoscopic Hysterectomy; Postoperative Recovery
Keywords: Intrathecal Morphine; Trocar-Site Infiltration; Intraperitoneal Bupivacaine; Laparoscopic Hysterectomy; Quality of Recovery (QoR-15); Postoperative Pain; Opioid Consumption; Inflammatory Markers; Neutrophil-to-Lymphocyte Ratio (NLR); Systemic Immune-Inflammation Index (SII)
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study uses a two-arm, parallel-group design in which participants are randomized in a 1:1 ratio to receive either intrathecal morphine or trocar-site plus intraperitoneal bupivacaine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This is a double-blind study. Participants and postoperative outcome assessors are blinded to group allocation. Randomization is generated by an independent researcher, and allocation is concealed in sequentially numbered opaque envelopes. The clinician performing the postoperative assessments is not involved in anesthesia administration and remains blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Morphine Group (Experimental): Participants in this arm will receive 200 µg of preservative-free intrathecal morphine administered at the L3-L4 interspace prior to induction of general anesthesia. This intervention is intended to provide early postoperative analgesia following laparoscopic hysterectomy.
  Interventions: Drug: Intrathecal Morphine
- Local Anesthesia Group (Active Comparator): Participants in this arm will receive 0.25% bupivacaine infiltration (5 mL at each trocar site) and 40 mL of 0.25% bupivacaine administered intraperitoneally at the end of surgery. The total dose of bupivacaine will not exceed 2 mg/kg. This technique aims to reduce postoperative somatic and visceral pain after laparoscopic hysterectomy.
  Interventions: Drug: Trocar-Site Bupivacaine Infiltration; Drug: Intraperitoneal Bupivacaine spray

INTERVENTIONS:
Drug: Intrathecal Morphine — A single dose of 200 µg preservative-free morphine will be administered intrathecally at the L3-L4 interspace prior to induction of general anesthesia. The injection is performed using a 25G spinal needle. This intervention aims to provide prolonged early postoperative analgesia in patients undergoing laparoscopic hysterectomy.
  Arms: Intrathecal Morphine Group
Drug: Trocar-Site Bupivacaine Infiltration — At the end of laparoscopic hysterectomy, 5 mL of 0.25% bupivacaine will be infiltrated into each trocar site. This intervention targets somatic pain originating from trocar entry points. It is administered only in the Local Anesthesia (LA) Group. The total dose of bupivacaine from all applications will remain within recommended safety limits.
  Arms: Local Anesthesia Group
Drug: Intraperitoneal Bupivacaine spray — A total of 40 mL of 0.25% bupivacaine will be instilled intraperitoneally after completion of the surgical procedure. This intervention is designed to reduce visceral and peritoneal irritation-related pain following laparoscopic hysterectomy. The combined bupivacaine dose from trocar-site infiltration and intraperitoneal instillation will not exceed 2 mg/kg.
  Arms: Local Anesthesia Group

SUMMARY:
This study aims to compare the effects of intrathecal morphine with trocar-site infiltration and intraperitoneal bupivacaine on postoperative pain control, quality of recovery, and inflammatory response in patients undergoing elective laparoscopic hysterectomy. Laparoscopic hysterectomy is widely used for benign gynecologic conditions, but postoperative pain may result from trocar-site trauma, peritoneal irritation, and carbon dioxide insufflation. Effective postoperative analgesia can improve patient comfort, reduce opioid use, and enhance early recovery.

Intrathecal morphine is known to provide potent early postoperative analgesia but may cause side effects such as nausea, vomiting, pruritus, and respiratory depression. Local anesthetic techniques, including trocar-site infiltration and intraperitoneal bupivacaine, have also been shown to reduce postoperative pain after minimally invasive gynecologic surgery.

In this prospective, randomized, double-blind study, patients will be assigned to one of two groups:

Intrathecal morphine (ITM) administered before induction of anesthesia;

Local anesthesia group (LA) receiving trocar-site infiltration and intraperitoneal bupivacaine at the end of surgery.

The primary outcome is the Quality of Recovery-15 (QoR-15) score at 24 hours. Secondary outcomes include pain scores, opioid consumption, time to first rescue analgesia, postoperative nausea and vomiting, pruritus, respiratory depression, early mobilization, bowel function recovery, and perioperative inflammatory markers such as neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), lymphocyte-to-monocyte ratio (LMR), and systemic immune-inflammation index (SII).

The results of this trial are expected to guide clinicians in selecting optimal analgesic strategies for laparoscopic hysterectomy and to contribute to improved patient recovery and postoperative satisfaction.

DETAILED DESCRIPTION:
Study Background and Rationale:

Despite its minimally invasive advantages, laparoscopic hysterectomy can cause significant postoperative pain due to trocar sites, visceral manipulation, and peritoneal irritation. This pain results in opioid consumption, associated side effects, and delayed recovery. Multimodal analgesia is the cornerstone of postoperative care. In this context, trocar site infiltration with intrathecal morphine (long-acting central analgesia) and intraperitoneal local anesthetic administration (peripheral techniques targeting somatic and visceral pain) are effective options. This study aims to compare the effects of these two different analgesic strategies on the quality of postoperative recovery through a patient-centered outcome measure, the QoR-15, and objective hematologic inflammatory markers.

Technical Details of Intervention Protocols:

General Anesthesia Standardization: All patients will receive standard general anesthesia. Induction will be achieved with propofol and fentanyl, rocuronium bromide will be used for neuromuscular blockade, and anesthesia will be maintained with sevoflurane.

Group ITM (Intrathecal Morphine) Intervention: Before induction of general anesthesia, patients will be in the sitting or lateral decubitus position and 200 µg (0.2 mg) of morphine will be injected into the subarachnoid space with a 25G (or 27G) pencil-point spinal needle at the L3-L4 intervertebral space. Hemodynamic and respiratory parameters will be closely monitored for 30 minutes after the injection.

Group LA (Local Anesthetic) Intervention: At the end of the surgical procedure, 5 mL of 0.25% bupivacaine will be infiltrated into each trocar incision. Additionally, 40 mL of 0.25% bupivacaine will be administered intraperitoneally, distributing to the subhepatic, diaphragmatic, and pelvic surfaces. The total bupivacaine dose will be calculated to avoid exceeding 2 mg/kg body weight to avoid the risk of toxicity.

Standard Perioperative Medication Regimen: All patients in both groups will receive the following medications intraoperatively as part of multimodal analgesia: 1 g Paracetamol, 800 mg Ibuprofen, 3 mg Granisetron, 40 mg Esomeprazole, and 8 mg Dexamethasone.

Methodological Details for Outcome Assessments:

QoR-15 Questionnaire: The validated and reliable Turkish version of the primary outcome measure, QoR-15, will be used. The questionnaire will be administered before surgery to obtain preoperative baseline values and at 24 hours postoperatively as the primary outcome.

Pain and Side Effect Monitoring: Postoperative pain will be assessed using a Visual Analog Scale (VAS: 0-10 cm) at rest and during coughing/activity. Assessments will be made at 2-hour intervals from the 2nd postoperative hour to the 24th hour. Nausea, vomiting, pruritus, and respiratory depression (SpO2 < 90% or respiratory rate < 8/minute) will be recorded using standard forms.

Hematological Inflammatory Markers: A complete blood count will be analyzed using an automated hematology analyzer from venous blood samples taken preoperatively (baseline, T0) and at the 24th postoperative hour (T13). Neutrophil/Lymphocyte Ratio (NLR), Platelet/Lymphocyte Ratio (PLR), Lymphocyte/Monocyte Ratio (LMR), and Systemic Immuno-Inflammation Index (SII = (Platelet count x Neutrophil count) / Lymphocyte count) will be calculated.

Blinding Protocol: Except for the anesthesiologist who performs the randomization and intervention, the patients, the surgical team, the investigators collecting postoperative data, and the statistical analyst will be blinded to group distinctions. Randomization will be stored using sequential, numbered, opaque envelopes.

Clinical Significance of the Study:

The findings of this study may provide evidence-based recommendations regarding the most effective multimodal analgesia regimen after laparoscopic hysterectomy. The demonstrated superiority of intrathecal morphine in reducing the systemic inflammatory response and patient-reported quality of recovery may result in less opioid use and faster recovery. Conversely, if local anesthetic techniques are adequate, the potential risks of central block may be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-65 years.
* Elective laparoscopic hysterectomy planned for benign gynecological conditions.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Ability to provide written informed consent.

Exclusion Criteria:

* Coagulopathy or bleeding disorders.
* Opioid dependence or chronic opioid use.
* Allergy or contraindication to local anesthetics or morphine.
* Contraindication to neuraxial (spinal) anesthesia.
* History of chronic pain syndromes.
* Severe renal or hepatic dysfunction.
* Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative quality of recovery at 24 hours measured by QoR-15 | 24 hours postoperatively
  The primary outcome is the overall postoperative recovery quality at 24 hours, assessed using the 15-item Quality of Recovery questionnaire (QoR-15). This scale evaluates physical comfort, emotional state, physical independence, psychological support, and pain to provide a comprehensive patient-centered measure of recovery.

SECONDARY OUTCOMES:
Time to first rescue opioid requirement | From end of surgery until first rescue opioid administration (up to 24 hours)
  Duration (in hours) from the end of surgery to the first administration of rescue opioid (oxycodone 5 mg) for postoperative pain relief.
Total opioid consumption within 24 hours | 0-24 hours postoperatively
  Total amount of rescue opioid consumed by the patient within the first 24 hours after surgery, expressed in milligrams.
Time to first mobilization | 0-24 hours postoperatively
  Time (in hours) from the end of surgery until the patient is able to ambulate independently for the first time postoperatively.
Time to first bowel movement | 0-24 hours postoperatively
  Time (in hours) from the end of surgery until the patient reports the first postoperative bowel movement.
Postoperative pain scores (VAS) | 2-24 hours postoperatively
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a continuous scale ranging from 0 to 10. Scores are recorded by patients marking a line, where 0 represents "no pain" and 10 represents "the worst pain imaginable". Higher scores indicate a worse outcome (more severe pain). Assessments will be performed at rest and during movement (e.g., coughing) at 2-hour intervals from 2 to 24 hours postoperatively.
Postoperative complications | 0-24 hours postoperatively
  Incidence of postoperative nausea, vomiting, pruritus, and respiratory depression within the first 24 hours after surgery.
Neutrophil-to-lymphocyte ratio (NLR) | Preoperative baseline and 24 hours postoperatively
  NLR measured preoperatively and at 24 hours postoperatively to evaluate systemic inflammatory response.
Platelet-to-lymphocyte ratio (PLR) | Preoperative baseline and 24 hours postoperatively
  PLR measured preoperatively and at 24 hours postoperatively to evaluate systemic inflammatory response.
Lymphocyte-to-monocyte ratio (LMR) | Preoperative baseline and 24 hours postoperatively
  LMR measured preoperatively and at 24 hours postoperatively to evaluate systemic inflammatory response.
Systemic immune-inflammation index (SII) | Preoperative baseline and 24 hours postoperatively
  SII measured preoperatively (T0) and at 24 hours postoperatively (T13) to evaluate systemic inflammatory response.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Dostbil, Principal Investigator, Principal Investigator — Ataturk University Department of Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive patient health information, and data confidentiality will be strictly maintained according to institutional ethical guidelines.

REFERENCES:
- [Background] Yang Y, Lin W, Zhuo Y, Luo Y, Wu X, Li J, Yao Y. Intrathecal Morphine and Ropivacaine for Quality of Recovery After Laparoscopic Colorectal Surgery: A Randomized Controlled Trial. Drug Des Devel Ther. 2024 Dec 18;18:6133-6143. doi: 10.2147/DDDT.S500316. eCollection 2024. PMID 39717198
- [Background] Xing H, Yuan D, Zhu Y, Jiang L. A nomogram model based on SII, AFR, and NLR to predict infectious complications of laparoscopic hysterectomy for cervical cancer. World J Surg Oncol. 2024 Jul 24;22(1):190. doi: 10.1186/s12957-024-03489-0. PMID 39049119
- [Background] Canikli Adiguzel S, Akyurt D, Bahadir Altun H, Tulgar S, Ultan Ozgen G. Can Neutrophil-Lymphocyte Ratio, Platelet-Lymphocyte Ratio, or Systemic Immune Inflammation Index Be an Indicator of Postoperative Pain in Patients Undergoing Laparoscopic Cholecystectomy? Cureus. 2023 Jan 19;15(1):e33955. doi: 10.7759/cureus.33955. eCollection 2023 Jan. PMID 36820108
- [Background] Aslanlar E, Aslanlar DA, Doganay C, Onal O, Sargin M, Cicekci F, Kara F, Kara I. The validity and reliability of the Turkish version of the quality of recovery-15 (QoR-15) questionnaire. Medicine (Baltimore). 2024 Apr 19;103(16):e37867. doi: 10.1097/MD.0000000000037867. PMID 38640327
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Pirie K, Doane MA, Riedel B, Myles PS. Analgesia for major laparoscopic abdominal surgery: a randomised feasibility trial using intrathecal morphine. Anaesthesia. 2022 Apr;77(4):428-437. doi: 10.1111/anae.15651. Epub 2022 Jan 17. PMID 35038165
- [Background] Kaya C, Dost B, Turunc E, Ustun YB, Kibar AN, Cebeci H, De Cassai A, Elsharkawy H. Unilateral subcostal anterior quadratus lumborum block versus intrathecal morphine for postoperative pain in laparoscopic nephrectomy: a randomized controlled trial. Reg Anesth Pain Med. 2025 Jul 10:rapm-2025-106844. doi: 10.1136/rapm-2025-106844. Online ahead of print. PMID 40639953
- [Background] Gluck O, Barber E, Feldstein O, Tal O, Kerner R, Keidar R, Wolfson I, Ginath S, Bar J, Sagiv R. The effect of subcutaneous and intraperitoneal anesthesia on post laparoscopic pain: a randomized controlled trial. Sci Rep. 2021 Jan 8;11(1):81. doi: 10.1038/s41598-020-80130-6. PMID 33420214
- [Background] Lirk P, Thiry J, Bonnet MP, Joshi GP, Bonnet F; PROSPECT Working Group. Pain management after laparoscopic hysterectomy: systematic review of literature and PROSPECT recommendations. Reg Anesth Pain Med. 2019 Apr;44(4):425-436. doi: 10.1136/rapm-2018-100024. Epub 2019 Feb 3. PMID 30914471
- [Background] Elsaeed UA, Algyoushy EAFIH, Hatem DLM. Effect of port-site and intraperitoneal local anesthetic injection versus placebo on postoperative pain and recovery after gynecologic laparoscopic surgery: a randomized controlled trial. Sci Rep. 2025 Sep 12;15(1):32466. doi: 10.1038/s41598-025-18389-w. PMID 40940430
- [Background] Antoun L, Smith P, Afifi Y, Cullis K, Clark TJ. Short stay laparoscopic hysterectomy: An evaluation of feasibility and patient satisfaction. Facts Views Vis Obgyn. 2021 Dec;13(4):377-385. doi: 10.52054/FVVO.13.4.039. PMID 35026099